CLINICAL TRIAL: NCT01567358
Title: A Randomized, Double-Blind, Repeated Dose, Active Control Drug, Parallel-group and Single-center Phase I Study of the Safety of Intravenous Administration of NI-071 in Comparison With Remicade® in Japanese Patients With Rheumatoid Arthritis Inadequately Treated With Methotrexate
Brief Title: Study of NI-071 in Comparison With Remicade in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nichi-Iko Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI071C1(ACT12719)
Record Dates: First submitted 2012-03-23; First posted 2012-03-30 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NI-071 (Experimental)
  Interventions: Biological: Infliximab
- Remicade (Active Comparator)
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — 100mg/vial
  Arms: NI-071
Biological: Infliximab — 100mg/vial
  Arms: Remicade

SUMMARY:
The purpose of this study is to compare the safety of NI-071 with Remicade® (infliximab) in patients with Rheumatoid Arthritis inadequately treated with Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Rheumatoid Arthritis (RA) as defined by the 1987 revised American College of Rheumatology (ACR) criteria with ACR Functional Classification class I-III and disease duration of no less than 3 months
2. Patients must receive a minimum of 3 months treatment with methotrexate (MTX) (≥ 6 mg/week) prior to the Screening Visit. Patients must be on a stable dose of MTX (6 mg~16 mg mg/week) for a minimum of 4 weeks prior to the Screening Visit

Exclusion Criteria:

1. History of following diseases

   * Other Connective tissue disorders with joint symptom which may interfere the efficacy assessment
   * Chlonic or recurrent infectious disease（bronchial ectasia, sinus inflammation etc.）
   * Severe infectious disease（hepatitis, pneumonia、sepsis）
   * History of demyelinating disease or multiple sclerosis
   * Congestive heart failure
   * lymphoproliferative disorder or myelodysplastic syndrome
   * History of malignancy
   * Interstitial lung disease
2. Patients with active or latent tuberculosis or history of tuberculosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety : Incidence of Adverse Events | 14 weeks

SECONDARY OUTCOMES:
PK : Area under the serum concentration versus time curve(AUC) | 14 weeks
Efficacy : ACR core-set | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 392001001, Sendai, Miyagi, Japan